CLINICAL TRIAL: NCT04601181
Title: A Study to Evaluate the Safety and Clinical Activity of Allogeneic CAR-T Targeting CD22 in Patients With Refractory or Relapsed B Cell Malignancies
Brief Title: Safety and Efficacy of ThisCART22 in Patients With Refractory or Relapsed B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundamenta Therapeutics, Ltd. (Industry)
Collaborators: The First Affiliated Hospital of USTC (Anhui Provincial Hospital) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART22
Record Dates: First submitted 2020-10-16; First posted 2020-10-23 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-10

CONDITIONS: B Cell Malignancy

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART22 cells injection (Experimental): In this arm，allogeneic anti-CD22 CAR T Cells(ThisCART22 cells) is used to treat patients with refractory or relapsed CD22 positive B cell malignancies.
  Interventions: Biological: ThisCART22 cells injection

INTERVENTIONS:
Biological: ThisCART22 cells injection — Assigned Interventions Biological/Vaccine: ThisCART22 cells 0.2-60 x 10^6 CAR-T cells per kg body weight.
  Intervention study

SUMMARY:
This is a single-center, nonrandomized, open-label, study to evaluate the safety and clinical activity of allogeneic CAR-T targeting CD22 in patients with refractory or relapsed CD22-positive B cell malignancies

DETAILED DESCRIPTION:
The patients will receive infusion of ThisCART22 cells from health donor ,to evaluate the safety and efficacy of ThisCART22 Cells in patients with refractory or relapsed CD22-positive B cell malignancies.

In this study, the dose range is 0.2-60 x10^6 cells per kg body weight (no more than 3.0 x 10^9 in total).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who volunteered to participate in the research and signed a written informed consent;
2. The informed consent was signed between the ages of 3-70, regardless of gender or race;
3. CD22 positive hematologic malignancies with no alternative treatment options deemed by investigator. including those who are not eligible for allogeneic stem cell transplantation (SCT) due to the following reasons： 3.1 age； 3.2 Concurrent disease； 3.3 Other contraindications, such as contraindications to total body irradiation (TBI) (TBI is one of the important treatment measures before allogeneic stem cell transplantation of ALL)； 3.4 Lack of suitable donors； 3.5 Patients with relapse after CD19-CAR T treatment；
4. Estimated life expectancy > 12 weeks deemed by investigator
5. Recurrence after any stem cell transplantation (regardless of previous treatment regimen);
6. Patients who relapse after previous allogeneic SCT (myeloablative or non-myeloablative) and meet all the following entry criteria:

   6.1 No active GVHD and no immunosuppression is required； 6.2 Transplant for more than 4 months；
7. Serum creatinine ≤1.6 mg/dl and/or BUN ≤ 1.5 mg/dl；
8. Serum ALT/ AST < 5 upper limit of normal (ULN)；
9. Measurable or detectable disease at time of enrollment，include minimal residual disease (MRD) detected by immunotyping, cytogenetics or PCR.
10. Cardiac ejection fraction ≥ 40%.
11. Eastern cooperative oncology group (ECOG) performance status of ≤ 2.
12. Female subjects with fertility have a negative pregnancy test result within 48 hours before the infusion and are not breast-feeding; all subjects with fertility potential before being enrolled in the study and throughout the study period until the last infusion Within 3 months, take adequate contraceptive measures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Participated in another clinical trial during the first 4 weeks of the enrolled study or intended to participate in another clinical trial throughout the study period;
3. Have been treated with any gene product;
4. Uncontrolled infection;
5. History of HIV infection;
6. Active hepatitis B virus or hepatitis C virus infection;
7. Systemic steroid therapy may be required for cell infusion or collection, or there may be conditions that the investigator considers may require steroid therapy during blood collection or infusion.Corticosteroids for disease treatment are permitted, and inhaled steroids or hydrocortisone physiologic replacement therapy for patients with adrenocortical dysfunction is permitted beyond the time of cell collection or infusion;
8. Patients with grade 2-4 GVHD, or deemed need to manage by investigator;
9. The presence of GVHD under treatment;.
10. Patients with active CNS involvement by malignancy;
11. Patients combine with other disease cause neutrophil count (ANC) <750/uL or PLT< 50,000/uL
12. The researchers considered the subjects unsuitable for this clinical trial for various reasons.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of AE or SAE of CART cell infusion in relation to the study drug at grade ≥3 (refer to CTCAE version 4.03); | From infusion to week 12
ORR (sum of CR and CRi) after infusion. | From infusion to week 12

SECONDARY OUTCOMES:
The survival time of CAR-T-22 cells in vivo; | From infusion to month 12
ORR at week 4, 8, and 24 after infusion (ORR4, ORR8, ORR24). | At week 4, 8, and 24 after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, M.D., Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No